CLINICAL TRIAL: NCT03511807
Title: Acoustic and Electrical Stimulation for the Treatment of Tinnitus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Hamid Djalilian, Professor, Otolaryngology, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20065187
Record Dates: First submitted 2018-02-01; First posted 2018-04-30 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Electricity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Electrical/ Acoustic stimulation (Experimental)
  Interventions: Other: Electrical; Other: Acoustic

INTERVENTIONS:
Other: Electrical — For the electrical stimulation:
  An electrode will be inserted into the ear canal which will be stimulated.
Other: Acoustic — For the acoustic stimulation:
  A typical sound will be presented for 6 minutes. Loudness is reported for 4 minutes after the stimulus offset to measure the presence and duration of the residual inhibition. If a successful acoustic stimulus is found, the subject will be given a series of sound files to listen to on a digital music player (CD or MP3 player) and will be asked to listen to each sound file (5 minute duration) and record their tinnitus loudness/annoyance during and after each sound stimulation. For some subjects, the investigators will use music on a digital music player (MP3 player) to see if music listening and music exercises will help reduce the intensity or annoyance level of the tinnitus (using the same surveys). These music-based exercises will involve training in recognition of musical intervals (e.g., octaves, fifths, and thirds).

SUMMARY:
Tinnitus, or ringing in the ears, affects 10% to 30% of the population. Of those, 20% have tinnitus bothersome enough to seek medical attention. In many people, tinnitus can significantly affect the quality of life. At this point in time, there is no effective treatment or cure available for tinnitus.

It has been found that electrical stimulation of the inner ear can reduce and in some cases eliminate tinnitus. The purpose of this research is to investigate both acoustic and electrical stimulation of the inner ear as a possible treatment of tinnitus.

In both acoustic and electrical testing conditions, the subjects will be instructed to be familiar with a 0-10 ranking scale of loudness. In acoustic testing, the stimulus will be presented through headphones in a noiseless environment, and the subject will be asked to report on the loudness of the presented sound and the level of the tinnitus at 20-second intervals. If the subject cannot perceive the presence of the tinnitus, a value of zero will be assigned. A typical sound will be presented for 3 to 6 minutes. Loudness will be reported for 1 to 4 minutes after stimulus offset to measure the presence and duration of residual inhibition.

Electrical stimulation will be delivered to the inner ear in three ways, 1. using a cochlear implant (implant placed in the inner ear to replace hearing function), 2. Using an electrode placed in the ear canal, and 3. using a small needle inserted through the ear drum. Various electrical signals will be used to evaluate the reduction in the tinnitus perception by the subject. The subjects will rate the loudness of the tinnitus before, during, and after the electrical signal. Surveys will be used to evaluate the tinnitus loudness and the quality of life of the subjects. Hearing tests will be used before and after the procedures. The long term goal of this research is to develop a device to treat tinnitus in people who can hear and to develop programs for cochlear implants that help treat tinnitus in deaf people.

DETAILED DESCRIPTION:
Tinnitus, or ringing in the ears, is a medical condition that significantly affects the quality of life of patients and that can be disabling to many. It has become known that acoustic and electrical stimulation of the inner ear can cause suppression and sometimes elimination of tinnitus. The long term goal of this study is to devise new methods for reduction/elimination of tinnitus. Multiple attempts at tinnitus suppression using acoustic and electrical stimulation of the inner ear has been performed with variable success. More commonly, acoustic stimulation is used to mask the tinnitus as opposed to suppressing or inhibiting the tinnitus. More recently, however, cochlear implants have been used for hearing as well as tinnitus suppression. The first hypothesis is that in using acoustic stimulation at specific frequencies and levels of loudness, tinnitus can be suppressed / eliminated. The second hypothesis is that using the same electrical stimulation technology as used in the cochlear implant, tinnitus can be suppressed/eliminated. These predictions will be tested in 3 specific aims. In Specific Aim 1, an acoustic sound will be delivered through headphones to the subjects' ears at various frequencies and loudness levels to evaluate suppression / elimination of tinnitus. In Specific Aim 2, an electrical current will be delivered to the inner ear. Pulse trains of various frequencies will be used to evaluate suppression/elimination of the ringing in the ears. Specific Aim 3. The effect of electrical stimulation on the subjects' quality of life will be measured using validated surveys.

In the past, attempts to suppress tinnitus using acoustic stimulation have succeeded in only masking the tinnitus to a limited degree. Tinnitus masking devices only camouflage the tinnitus. Patients frequently report an interference with hearing or complain that the devices only substitute one unpleasant sound for another. Additionally, the masking devices can only be used for a limited time and the patient's tinnitus often subjectively becomes worse after the removal of the device. Patients also become habituated or accustomed to the device thereby decreasing its effectiveness over time.

Attempts to suppress tinnitus using electrical stimulation have a long history. Starting in 1801 and continuing throughout the 19th century, the effects of electrical stimulation on the ear were described by several authors. Some of these early attempts showed that direct current applied to the mastoid or zygoma could suppress and possibly eliminate tinnitus in some patients. Aran et al have found that electrical stimulation of the inner ear via an electrode inserted through the ear drum can cause suppression and sometimes elimination of tinnitus.

The advent of the cochlear implant revolutionized the restoration of hearing to the deaf by electrically stimulating the hearing nerve. As a side-benefit, the cochlear implant was found to suppress tinnitus in 28% to 79% of patients. Electrical stimulation of the inner ear may have a direct electrical influence on the tinnitus generated in the inner ear, or it may have an indirect influence by creating activity centrally where tinnitus reduction occurs. The success with cochlear implants has led to a number of studies to evaluate electrical stimulation for suppression of tinnitus. These studies have used electrodes externally and internally (behind the ear drum) and various stimulus waveforms. They all suggest that in some patients, tinnitus can be suppressed and occasionally eliminated using these techniques. It is important to note that none of these studies was placebo-controlled.

Most recently in a preliminary study in 2003, Rubinstein et al, used a needle electrode passed through the ear drum to suppress tinnitus. The authors used a high pulse rate of 4,800 pulse-per- second (pps) for their electrical stimulation. They found that 5 of 11 (45%) subjects with electrical stimulation of the inner ear through the ear drum using a needle electrode showed substantial or complete tinnitus suppression with either no perception or only a transient perception of the stimulus. Three (27%) showed tinnitus suppression with the perception of the stimulus and three showed no suppression of the tinnitus. In subjects with cochlear implants, the authors used the cochlear implant for tinnitus suppression using the electrical signal sent through the implant to the inner ear. The results of tinnitus suppression using the cochlear implant were similar to the subjects without implants. Based on recent work performed on cochlear implant subjects, it has been found that low pulse rate stimulation may be more beneficial in suppressing tinnitus in cochlear implant patients. Electric stimulation will be delivered through an optically-isolated constant-current source. The maximum output will be set at 1000 microamps and be periodically calibrated to ensure accuracy. This device has been used in several previous studies on hearing perception and a similar device has been used to treat tinnitus . The device is routinely used for cochlear implant patients, but is not routinely used to stimulate people without cochlear implants (given their normal hearing status). It has been used experimentally, however, used for people with hearing loss or tinnitus.

The goal of this study is to expand on these studies and to evaluate the impact of various modes of electrical stimulation for the suppression of tinnitus and to evaluate the quality of life impact of tinnitus suppression on the patients. The predictor variables include frequency, pulse width, and waveform of the electrical stimulation. This study will determine which combination of amplitude, frequency, or waveform will provide the best response. If successful, this method of treating tinnitus could form the basis for development of hopefully the first effective treatment for tinnitus.

The outcome variables include tinnitus level (on a scale of 0-100, with 100 being the loudest level of tinnitus they have experienced), tinnitus handicap inventory score, and Short-form 36 results.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Male or female
3. Tinnitus present for 6 months or more
4. Adequate command of English to reliably describe the unusual sensory percepts provided by electrical stimulation, and to complete surveys.
5. For patients undergoing electrical stimulation via a cochlear implant, they should have a cochlear implant prior to enrollment (not applicable for acoustic stimulation)

Exclusion Criteria:

1. Aged less than 18 years
2. Active illicit drug use, alcohol dependence
3. Treatable cause of tinnitus
4. History of psychosis
5. Abnormalities of the ear canal or ear drum
6. Chronic middle ear disease
7. Subjects on medications known to cause tinnitus (aspirin, ibuprofen, naproxen) which could not be stopped will be excluded.
8. Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Audiogram | Occurs once at the beginning of subject participation (less than one hour)
  Measures hearing ability in db hearing loss (HL).
Otoacoustic Emissions (OAE) | Occurs once at the beginning of subject participation (less than one hour)
  Measures health of the inner ear in db hearing loss (HL).
Tinnitus Handicap Inventory (THI) | Outcome will be measured during each participant visit through study completion which can be an average of 1 year
  Quantifies and evaluates difficulties experience because of tinnitus measured in a numerical score range: Yes (value of 4, highest) Sometimes (value of 2) and No (value of 0, lowest). The sum of all responses yields a total THI score (0-100). High scores indicate catastrophic handicap. Low scores indicate slight or no handicap.
Medical Outcomes Study Questionnaire Short Form 36 (SF-36) Health Survey Quality of life metrics. | Outcome will be measured during each participant visit through study completion which can be an average of 1 year
  The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0-100. Lower scores indicate more disability, higher scores indicate less disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Hamid R. Djalilian, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feldman H. History of tinnitus research. In: Shulman A, ed. Tinnitus Diagnosis/Treatment. San Diego: Singular Publishing Group; 1997:3-37.
- [Background] de Sauvage RC, Cazals Y, Aran JM. Observation of an electrically evoked whole-nerve response using the same stimulating and recording electrode: an image of the unit response at the round window (preliminary report). Hear Res. 1980 Jun;2(3-4):343-6. doi: 10.1016/0378-5955(80)90068-4. No abstract available. PMID 7410238
- [Background] Zwolan TA, Kileny PR, Souliere CR, Kemink JL. Tinnitus suppression following cochlear implantation. In: Aran J-M, Dauman R, eds. Tinnitus 91: Proceedings of the Fourth International Tinnitus Seminar. Amsterdam: Kugler, 1992;423-6.
- [Background] Rubinstein JT, Tyler RS, Johnson A, Brown CJ. Electrical suppression of tinnitus with high-rate pulse trains. Otol Neurotol. 2003 May;24(3):478-85. doi: 10.1097/00129492-200305000-00021. PMID 12806303
- [Background] Kuk FK, Tyler RS, Rustad N, Harker LA, Tye-Murray N. Alternating current at the eardrum for tinnitus reduction. J Speech Hear Res. 1989 Jun;32(2):393-400. doi: 10.1044/jshr.3202.393. PMID 2786979
- [Background] Hazell JW, Jastreboff PJ, Meerton LE, Conway MJ. Electrical tinnitus suppression: frequency dependence of effects. Audiology. 1993;32(1):68-77. doi: 10.3109/00206099309072929. PMID 8447763
- [Background] Okusa M, Shiraishi T, Kubo T, Matsunaga T. Tinnitus suppression by electrical promontory stimulation in sensorineural deaf patients. Acta Otolaryngol Suppl. 1993;501:54-8. doi: 10.3109/00016489309126215. PMID 8447227
- [Background] Ito J, Sakakihara J. Tinnitus suppression by electrical stimulation of the cochlear wall and by cochlear implantation. Laryngoscope. 1994 Jun;104(6 Pt 1):752-4. doi: 10.1288/00005537-199406000-00017. PMID 8196452
- [Background] Matsushima JI, Sakai N, Uemi N, Miyoshi S, Sakajiri M, Ifukube T. Evaluation of Implanted Tinnitus Suppressor Based on Tinnitus Stress Test. Int Tinnitus J. 1997;3(2):123-131. PMID 10753374
- [Background] Shulman A. External electrical stimulation in tinnitus control. Am J Otol. 1985 Jan;6(1):110-5. No abstract available. PMID 3872077
- [Background] Vurek LS, White M, Fong M, Walsh SM. Opto-isolated stimulators used for electrically evoked BSER: some observations on electrical artifact. Ann Otol Rhinol Laryngol Suppl. 1981 Mar-Apr;90(2 Pt 3):21-4. doi: 10.1177/00034894810902s208. No abstract available. PMID 6784647
- [Background] Zeng FG, Shannon RV. Loudness-coding mechanisms inferred from electric stimulation of the human auditory system. Science. 1994 Apr 22;264(5158):564-6. doi: 10.1126/science.8160013.